CLINICAL TRIAL: NCT02401126
Title: Dietary Nitrate Supplementation and Cardiorespiratory Control in Chronic Heart Failure: a Randomized, Placebo-controlled Trial
Brief Title: Effects of Dietary Nitrate Supplementation on Cardiorespiratory Control in Chronic Heart Failure
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Queen's University (Other)
Responsible Party: Principal Investigator, Dr. J. Alberto Neder, Principal Investigator, Queen's University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 6012610
Record Dates: First submitted 2015-03-24; First posted 2015-03-27 (Estimated); Last update posted 2016-05-02 (Estimated); Status verified 2016-04

CONDITIONS: Heart Failure, Systolic
MeSH Terms: conditions — Heart Failure, Systolic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nitrate supplementation (Active Comparator): Concentrated nitrate-rich beetroot juice
  Interventions: Dietary Supplement: Nitrate supplementation
- Placebo (Placebo Comparator): Nitrate-depleted beetroot juice
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Nitrate supplementation — Nitrate supplementation: concentrated nitrate-rich beetroot juice (2 x 70 ml/day; approximately 10 mmol nitrate/day; Beet It, James White Drinks, Ipswich, UK) for 8 consecutive days.
  Other Names: Concentrated nitrate-rich beetroot juice
  Arms: Nitrate supplementation
Dietary Supplement: Placebo — Placebo: nitrate-depleted beetroot juice (2 x 70 ml/day; approximately 0.01 mmol nitrate/day; Beet It, James White Drinks, Ipswich, UK) for 8 consecutive days. The placebo juice is similar to the concentrated beetroot juice in appearance, texture, smell and taste and is obtained by removing nitrate ions from the latter.
  Other Names: Nitrate-depleted beetroot juice
  Arms: Placebo

SUMMARY:
The main purpose of this study is to determine whether dietary nitrate supplementation via concentrated beetroot juice improves central and peripheral cardiovascular control and physical capacity in patients with systolic heart failure.

DETAILED DESCRIPTION:
Chronic heart failure (CHF) is a leading cause of morbidity and mortality worldwide. Although affecting the heart at first, it is now recognized that disability is largely due to impaired cerebral and skeletal muscle blood flow and consequently microvascular oxygenation. Reduced muscle oxygenation compromises oxidative metabolism and thus contractile performance. Impaired cerebral oxygenation not only reduces motor output (thus exacerbating muscle fatigue) but also constitutes a predictor of cerebral ischemic events and an independent prognostic risk factor.

Reduced levels of the vasodilator nitric oxide (NO) contribute to impaired blood flow and oxygenation in CHF. Development of new effective therapeutic strategies is therefore crucial given that current pharmacological treatment has failed to abrogate oxygenation deficits in CHF patients. Emerging evidence shows that nitrate serves as an alternative source for NO and improves muscle blood flow and oxygenation in health. Another striking feature of nitrate is that it can improve muscle work efficiency, a tenet of physiology that was once considered immutable.

Objective: To investigate systematically the role of dietary nitrate supplementation on central and peripheral cardiovascular function in CHF patients.

ELIGIBILITY:
Inclusion Criteria:

- previous diagnosis of systolic heart failure (left ventricular ejection fraction <40%) under optimized clinical treatment as judged by the accompanying physician.

Exclusion Criteria:

* hospital admission in the previous 6 weeks;
* exercise training program in the previous 6 months;
* nitrate therapy (e.g., isosorbide dinitrate);
* tabagism;
* any condition that could interfere with the ability to exercise;
* diagnosed psychiatric or cognitive disorders;
* type I insulin-dependent diabetes mellitus;
* excessively over-weight (BMI>35kg/m²);
* other diagnosed cardiorespiratory disorders (e.g., chronic obstructive pulmonary disease, peripheral artery disease).

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2015-03; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Exercise tolerance | 8 days
  Cycle ergometer exercise test to the limit of tolerance

SECONDARY OUTCOMES:
Plasma nitrate and nitrite concentrations | 8 days
  Assessed by chemiluminescence
Central and peripheral fatigue | 8 days
  Assessed by transcutaneous femoral nerve magnetic stimulation
Skeletal muscle and cerebral blood flow and oxygenation | 8 days
  Assessed by near-infrared spectroscopy and the rate of appearance of the optically-dense indocyanine green dye
Neuromuscular activity | 8 days
  Assessed by electromyography
Dyspnea and leg effort scores | 8 days
  Evaluated via a 10-point Borg scale
Cognitive performance | 8 days
  Assessed by computer-based tests
Cardiorespiratory responses to exercise | 8 days
  Non-invasive evaluation of cardiac (mean arterial pressure, cardiac output, stroke volume and heart rate) and pulmonary gas exchange (e.g., minute ventilation and oxygen uptake) responses during the transition from rest to exercise

CONTACTS AND LOCATIONS:
Overall Officials: J. Alberto Neder, MD, PhD, Principal Investigator — Queen's University